CLINICAL TRIAL: NCT01578538
Title: Mesh Used Repairs in Emergency Abdominal Wall Hernias
Brief Title: Safety of Mesh Used Repairs in Emergency Abdominal Wall Hernias. Prospective Randomized Multicenter Trial
Acronym: hernia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: SB Istanbul Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Erhan Aysan, prof. dr., SB Istanbul Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: herni; travma & emergency surgery (Registry Identifier: mcs)
Record Dates: First submitted 2012-04-13; First posted 2012-04-17 (Estimated); Last update posted 2012-04-17 (Estimated); Status verified 2012-04

CONDITIONS: Hernia
Keywords: hernia, abdominal, strangulation, emergency, wall
MeSH Terms: conditions — Hernia; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- mesh used repair (Active Comparator): mesh used hernia repair will be perform
  Interventions: Procedure: inguinal hernia repair
- nonmesh (Active Comparator): nonmesh hernia repair techniques will be used
  Interventions: Procedure: inguinal hernia repair

INTERVENTIONS:
Procedure: inguinal hernia repair — strangulated hernias will be repaired surgically

SUMMARY:
Repairing of emergency (strangulated) abdominal wall hernias with mesh may cause infective complications.

DETAILED DESCRIPTION:
Repairing of emergency (strangulated) abdominal wall hernias with mesh is controversary. Strangulated abdominal hernias are not clean surgical wounds so applying prostetic materials such as meshes are problematic. Using of prostetic materials in un-clean wounds (clean contaminated, contaminated and dirty) is not proposed. But in surgical practice meshed surgical repair techniques are using largeley. In this multicenter study we try to find the answer for emergency hernia repairs meshed or not.

ELIGIBILITY:
Inclusion Criteria:

1. Older than 16 years old,
2. Strangulated abdominal wall hernia
3. No any contrindications to operation

Exclusion Criteria:

1. Younger than 16 years old,
2. Non-strangulated abdominal wall hernis
3. Any causes of contrindications to operation

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-02; Primary Completion 2014-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
wound infection | six months
  surgical wound infection is the primary outcome measure of this trial

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University, Istanbul, Marmara, Turkey (Türkiye)